CLINICAL TRIAL: NCT06009419
Title: Effectiveness of Dual Task Training Versus Usual Care in Patients With Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Effectiveness of Dual Task Training in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kalça artroplasti dualtask
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Hip Arthroplasty
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the program given to the control group, the dual task program will be progressively given to the study group as previously described (Silsupadol et al., 2006). These applications will be explained to the patients or their relatives face-to-face in the clinical environment after the initial evaluation and then sent and followed up by telerehabilitation method and patients will always have access to programs and education. In addition, both groups will be told that they can contact the researcher upon request.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive the usual post-operative care of stretching lower extremity strengthening balance exercises activities of daily living recommendations.
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The control group will receive the usual post-operative care of stretching, lower extremity strengthening, balance exercises, activities of daily living recommendations. The study group will be given a dual task program in addition to the program given to the control group.

SUMMARY:
This study was planned to investigate the effectiveness of usual care and dual task program in patients who underwent total hip arthroplasty surgery. It is aimed to evaluate pain intensity, disability level, mini mental status, coordination, balance and functional status of the patients. The study will be conducted with volunteer patients who are followed up by the Orthopedics and Traumatology outpatient clinic of Muğla Training and Research Hospital and who have undergone total hip arthroplasty surgery. The evaluations will be performed in the Orthopedics and Traumatology outpatient clinic of Muğla Training and Research Hospital. It is aimed to evaluate at least 24 patients for the study.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone unilateral total hip arthroplasty surgery and being 6 weeks postoperative
* Participate in all necessary follow-up assessments
* 60 years of age or older
* Understand simple commands
* Signing the consent form

Exclusion Criteria:

* A previous history of total hip arthroplasty
* Presence of revision surgery
* Presence of severe osteoarthritis in the contralateral hip
* Severe acute metabolic neuromuscular and cardiovascular diseases
* Severe obesity (bki>35)
* Presence of malignancy
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that prevent communication
* Lack of cooperation during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Five Times Sit to Stand Test (5TSST) | Change from Baseline 5TSST at 8 weeks
  A chair without armrests, with a 28.5 cm deep seat and backrest and adjustable height is used for the tests. Subjects start in a seated position, with their arms in the desired position and their backs against the chair backrest. The following verbal instructions are given: "Please stand up and sit down 5 times as quickly as possible. Straighten your knees when standing up and lean your back against the backrest when sitting down." Timing with the digital stopwatch is started manually with the instruction "Start" and stopped when the subject's back touches the backrest after the fifth standing up.
Cognitive Timed Up and Go Test (CTUG) | Change from Baseline CTUG at 8 weeks
  Patients are first asked to stand up from a sitting position, walk 3 m at their normal speed, turn around, walk back to the chair and sit down. Walking aids are allowed. Patients are asked to perform this test while performing a cognitive dual task (subtract 2 continuously starting from 100).
Dual-Task Questionnaire (DTQ) | Change from Baseline DTQ at 8 weeks
  The questionnaire consists of 10 items and each question is rated out of 5 points (ranging from 0 "never" to 4 "very often" or N/A "not applicable"). The score obtained is the average score per question (i.e. total score/10 for the questionnaire).
Activity Specific Balance Confidence Scale (ABC) | Change from Baseline ABC at 8 weeks
  This scale includes 16 tasks related to indoor and outdoor activities of daily living to measure balance confidence in older people with various levels of function. Scores for each question range from 0% (no confidence) to 100% (full confidence). Higher scores indicate greater confidence.
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 10 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
Harris Hip Score (HHS) | Change from Baseline HHS at 8 weeks
  The HHS contains 12 questions covering four domains: pain (44 points); function (47 points); deformity; and range of motion (9 points). This questionnaire was developed to assess the outcomes of young and middle-aged patients following hip arthroscopic debridement. Each question is answered using a Likert scale with an overall score ranging from 0 (extreme symptoms) to 100 (no symptoms).
Mini-Mental State Examination (MMSE) | Change from Baseline MMSE at 8 weeks
  The mini mental test is categorized under five main headings: orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). The scale is scored out of a total of 30 points and has two different variants for educated and uneducated people. Traditionally, scores between 24 and 30 are considered normal. A score below 24 indicates cognitive impairment. 18-23 is considered as mild dementia, 12-17 as moderate dementia and below 12 as severe dementia.
Lower-Extremity Motor Coordination Test (LEMOCOT) | Change from Baseline LEMOCOT at 8 weeks
  The test requires subjects seated in a chair to alternately touch a proximal and distal target placed 30 cm apart on the floor with their feet within a 20-second period. A higher score indicates better motor coordination.
4-Meter Gait Speed (4MGS) | Change from Baseline 4MGS at 8 weeks
  Walking speed is assessed over two trials using a stopwatch in a long corridor over a distance of 4 meters during a single testing session, with one trial performed immediately after the other. Participants start ambulating approximately two meters before the start of the timed 4-meter walk and stop ambulating approximately two meters after completing the 4-meter walk. Timing begins and ends when the participants' lead foot crosses the start and end points of the 4-meter walk, respectively. Participants are instructed to walk at their normal safe walking speed and are allowed to use an assistive device if needed. The time taken to complete the two ambulation trials is recorded for analysis. Walking speed is calculated as the distance walked (4 meters) divided by the time taken to complete the 4-meter walk. The average walking speed for the two trials is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Uysal I, Ozden F, Yalcin M, Isik EI, Sari Z. The effect of dual-task training in older adults with total hip arthroplasty: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Jan 8;26(1):29. doi: 10.1186/s12891-025-08279-7. PMID 39780083